CLINICAL TRIAL: NCT03197077
Title: A Comparison Between Corifollitropin Alfa and Recombinant FSH for Follicular Recruitment in Women With Polycystic Ovaries Who Undergo IVM Treatment
Brief Title: Optimisation of Follicular Recruitment in IVM Cycles
Acronym: Elonva_IVM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Michel De Vos, Medical director, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017.corifollitropinalfa_IVM
Record Dates: First submitted 2017-06-16; First posted 2017-06-23 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Infertility, Female; Polycystic Ovary Syndrome
MeSH Terms: conditions — Infertility, Female; Polycystic Ovary Syndrome | interventions — Blood Specimen Collection; Oocyte Retrieval; Intravital Microscopy; follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta; Contraceptives, Oral; Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elonva (Experimental): A single injection of 100 microgram corifollitropin alfa. Oocyte retrieval on day five after corifollitropin alfa injection.
  Interventions: Procedure: blood sampling; Procedure: transvaginal ultrasound scanning; Procedure: oocyte retrieval for IVM; Drug: Corifollitropin Alfa; Drug: oral contraceptive pill pretreatment (Marvelon)
- Puregon (Active Comparator): Three daily injections of 150 IU follitropin beta. Oocyte retrieval on day five after the first follitropin beta injection.
  Interventions: Procedure: blood sampling; Procedure: transvaginal ultrasound scanning; Procedure: oocyte retrieval for IVM; Drug: Follitropin beta; Drug: oral contraceptive pill pretreatment (Marvelon)

INTERVENTIONS:
Procedure: blood sampling — comparison between corifollitropin alfa and follitropin beta in IVM cycles
Procedure: transvaginal ultrasound scanning — comparison between corifollitropin alfa and follitropin beta in IVM cycles
Procedure: oocyte retrieval for IVM — comparison between corifollitropin alfa and follitropin beta in IVM cycles
Drug: Corifollitropin Alfa — Single injection of 100 micrograms of corifollitropin alfa
  Arms: Elonva
Drug: Follitropin beta — Daily injection (three days) of follitropin beta
  Arms: Puregon
Drug: oral contraceptive pill pretreatment (Marvelon) — Daily administration of the oral contraceptive pill (Marvelon) for 21 days. Administration of the combined oral contraceptive pill will start after a blood test that demonstrates basal E2 levels and a negative serum hCG level.

SUMMARY:
The study will focus on important aspects related to follicle recruitment using exogenous gonadotropins in patients with polycystic ovaries:

1. Early follicle recruitment in patients with polycystic ovaries using corifollitropin alfa: does administration of this drug result in earlier and higher FSH (follicle stimulating hormone) concentrations above the threshold for follicle recruitment in an IVM (in vitro maturation) cycle preceded by oral contraceptive suppression, in comparison to normal daily administration of rFSH (recombinant follicle stimulating hormone, Puregon)?;
2. The maturation rate of the obtained oocyte-cumulus complexes in standard IVM media registered for clinical use: does stimulation with corifollitropin alfa versus recombinant FSH have an impact on the maturation rate and developmental capacity of the oocytes ?

ELIGIBILITY:
Inclusion Criteria:

1. Subfertile patients between 18-36 years old eligible for ART treatment
2. BMI 18-30
3. Polycystic ovaries (PCO) according to the Rotterdam criteria (at least 12 antral follicles per ovary as observed on a baseline ultrasound scan), with or without hyperandrogenism, with or without oligoamenorrhoea. In other words, patients are eligible if they have PCO morphology. A diagnosis of PCOS (polycystic ovary syndrome) based on Rotterdam criteria is not compulsory.

Exclusion Criteria:

1. Antral follicle count (AFC) <24
2. Anti-müllerian hormone (AMH) <3,25 in non-OCP (oral contraceptive pill) users and <4,00 in current OCP users (using Elecsys platform (Roche Diagnostics))
3. Couples requesting PGD (preimplantation genetic diagnosis)
4. Non-obstructive azoospermia in the male partner

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of COC | 5 days after the first gonadotropin injection (on the day of oocyte retrieval)
  Number of oocyte cumulus complexes obtained on the day of oocyte retrieval.

SECONDARY OUTCOMES:
Clinical pregnancy rate | At about 6 - 7 weeks gestation
  Clinical pregnancy rate after the first embryo transfer following the IVM cycle

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No